CLINICAL TRIAL: NCT02001376
Title: A Health Promotion Project for Workers at National Taiwan University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 201007040R
Record Dates: First submitted 2013-09-25; First posted 2013-12-04 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-08

CONDITIONS: Abdominal Obesity Metabolic Syndrome; Subjects With Poor Fitness Status
MeSH Terms: conditions — Abdominal obesity metabolic syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intensive exercise & home exercise (Experimental): Intensive exercise group Home exercise group
  Interventions: Other: Intensive exercise; Other: Home exercise
- Intensive exercise & control (Experimental): Intensive exercise group Control group
  Interventions: Other: Intensive exercise; Other: Control group live as usual
- Home exercise & control group (Experimental): Home exercise Control group
  Interventions: Other: Home exercise; Other: Control group live as usual

INTERVENTIONS:
Other: Intensive exercise — The intensive exercise group will receive moderate aerobic exercise and strengthening exercise three times a week for three months.
  Arms: Intensive exercise & control; Intensive exercise & home exercise
Other: Home exercise — The home-based exercise group will receive exercise instruction biweekly for three months
  Arms: Home exercise & control group; Intensive exercise & home exercise
Other: Control group live as usual — Control group means no any intervention for them. The control group who with metabolic syndrome risk factors just live as usual.
  Other Names: Control group
  Arms: Home exercise & control group; Intensive exercise & control

SUMMARY:
Background and Purpose: Fitness is the foundation for health and quality of life for individuals. Recent changes in lifestyle and eating habit in Taiwan have significantly increased the prevalence of metabolic syndrome that may lead to poor fitness and subsequent coronary artery disease, cardiovascular disease and diabetes. Although workers at the National Taiwan University Hospital (NTUH) have undertaken regular health fitness examination, the examination did not include the posture and movement analysis and no exercise intervention was provided to those with metabolic syndrome. This study is therefore aimed to conduct comprehensive health fitness examination for workers at NTUH and to examine whether exercise intervention could decrease the risk factors and enhance fitness in those at risk or with metabolic syndrome. Methods: This study will consist of two parts. In the first part, 1102 workers at NTUH will be administered comprehensive fitness examination (body mass index, waist circumference, muscle strength, flexibility, balance, cardiopulmonary test, and posture and movement analysis) and will be assessed with the Physical Activity Readiness and the Perceived Musculoskeletal Pain Scale and the International Physical Activity Questionnaire. Those workers who are at risk or have metabolic syndrome (N=240) will be assigned into the control, home-based exercise, and intensive exercise group with 80 in each group with their will. The home-based exercise group will receive exercise instruction biweekly for three months; the intensive exercise group will receive moderate aerobic exercise and strengthening exercise three times a week for three months. The other workers who are insufficient fitness status (N=240) will be assigned into the control, home-based exercise, and intensive exercise group with their will. The home-based exercise group will receive exercise instruction biweekly for a month; the intensive exercise group with 80 in each group will receive moderate aerobic exercise and strengthening exercise three times a week for a month. Descriptive statistics will be used to estimate the prevalence of 1, 2 and ≧3 metabolic risk factors, and poor fitness. One-way analysis of variance (ANOVA) will be used to examine the relation between metabolic syndrome risk factors and fitness. One-way ANOVA will be used to compare the demographic characteristics of the control, home-based exercise, and intensive exercise group. Two-way ANOVA repeated measures will be used to examine the metabolic syndrome risk factors and fitness in the three groups across time. Clinical relevance: Our results will help understand the health fitness of workers at NTUH and will assist in establishing effective exercise program for those at risk or with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-60 years old
* At least one metabolic syndrome risk factor (Elevated blood pressure: Equal to or greater than 120/80 mm Hg, Central obesity: waist circumference ≥ 90 cm (male), ≥ 80 cm (female), Elevated triglycerides: Equal to or greater than 150 mg/dL, Reduced HDL cholesterol: Men - Less than 40 mg/dL Women - Less than 50 mg/dL, Elevated fasting glucose: Equal to or greater than 100 mg/dL)

Exclusion Criteria:

* diastolic blood pressure greater than 139 mm Hg or systolic blood pressure greater than 89 mm Hg
* fasting glucose greater than 125 mg/dL
* triglycerides greater than 199 mg/dL
* Subjects have in progress cardiovascular disease or in treatment course
* chest distress, short of breath, dizziness, faint in recent 3 months
* Muscular skeletal system injury or pain

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-04; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
All improve fitness status | 36 weeks
  Body mass index, BMI is calculated by dividing a person's weight (in kilograms) by his or her height (in meters, squared).

SECONDARY OUTCOMES:
All improve fitness status | 36 weeks
  waist circumference To measure waist circumference locate the top of the hip bone. Place the tape measure evenly around the bare abdomen at the level of this bone. Read the tape measure and record the waist circumference in centimeters.
  The following individuals are at increased risk for developing chronic diseases:
  Women with a waist circumference of more than 80 centimeters. Men with a waist circumference of more than 90 centimeters.

OTHER OUTCOMES:
All improve fitness status | 36 weeks
  muscle strength The Curl-Up Test is to assess the endurance of the subjects' abdominal muscles.
All improve fitness status | 36 weeks
  muscle flexibility The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles.
All improve fitness status | 36 weeks
  balance One leg standing with eye-closed, assess bilateral legs.
All improve fitness status | 36 weeks
  cardiopulmonary index The 3-Minute Step Test measures subjects' aerobic (cardiovascular) fitness level based on how quickly subjects' heart rate returns to normal after exercise.
All improve fitness status | 36 weeks
  posture and movement analysis Posture is more than how subject look when sitting or standing. Good posture is defined as the ideal spine alignment and body positioning that puts the least strain on the body. Good posture distribute weight and forces evenly so that no one body region is overstressed. Good posture reduces the stress on joints, protects the ligaments supporting the spine, and allows muscles to work efficiently to reduce fatigue. Bad posture puts abnormal stress on the spine and can cause premature development of conditions such as spine arthritis and degenerative disc disease. Good posture put the weight line straight along ear, acromial and great trochanter.

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Physical Therapy Center, National Taiwan University Hospital, Taipei, Taiwan